Created on: 16.04.2024

## INFORMED CONSENT FORM

Study Title: Prevalence of Sexual Dysfunction in Female Patients with Multiple Sclerosis and Its Relationship with Various Factors

You are invited to participate in this study. Before you decide, it is important that you understand why the research is being done and what it will involve. Please read the following information carefully and ask any questions you may have.

## Purpose of the Study:

The aim of this study is to determine the prevalence of sexual dysfunction in female patients diagnosed with multiple sclerosis and to evaluate its relationship with fatigue, depression, anxiety, cognitive dysfunction, and overactive bladder symptoms.

#### Procedures:

If you agree to participate, you will be asked to complete the following questionnaires:

- Female Sexual Function Index (FSFI)
- Brief International Cognitive Assessment for MS (BICAMS)
- Hospital Anxiety and Depression Scale (HADS)
- Fatigue Severity Scale (FSS)
- Overactive Bladder Questionnaire (OAB-V8)

Completion of these questionnaires is expected to take approximately 60-90 minutes.

# Number of Participants:

Approximately 140 volunteers are expected to participate.

#### Potential Benefits and Risks:

There is no anticipated harm in participating in this study. The results may help improve the quality of life and contribute to scientific knowledge.

# Confidentiality:

All personal and medical information will remain confidential and will only be used for scientific purposes. Your identity will not be revealed in any reports or publications.

## Voluntary Participation and Withdrawal:

Your participation is voluntary. You may withdraw from the study at any time without penalty or loss of rights.

# Responsible Investigator:

Name: Merve Dokumaci

Affiliation: Ege University Faculty of Medicine, Department of Physical Medicine and Rehabilitation

Phone: +90 543 508 8428

#### **Consent Statement:**

I have read and understood the information provided above. I have had the opportunity to ask questions and all my questions have been answered. I voluntarily agree to participate in this study. I understand that I will receive a signed and dated copy of this informed consent form.

| Participant's Name and Signature: _ | Date: |
|-------------------------------------|-------|
| Researcher's Name and Signature: | Date: |